CLINICAL TRIAL: NCT02003950
Title: Effect of Three-Week Chocolate Candy Restriction on Pre- and Post-restriction Chocolate Candy Consumption in Healthy Adults
Brief Title: Pre- and Post-restriction Chocolate Candy Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Professor, Food and Nutrition, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 055-037; 0911008653 (Registry Identifier: Purdue University)
Record Dates: First submitted 2013-11-15; First posted 2013-12-06 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Investigate the Maladaptive Eating Behaviors of Normal Healthy Adults

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Chocolate pre-restriction (Other)
  Interventions: Other: Snack Condition Specification
- Chocolate Baseline (Other)
  Interventions: Other: Snack Condition Specification
- Chocolate post-restriction (Other)
  Interventions: Other: Snack Condition Specification
- Salty Snacks (Other)
  Interventions: Other: Snack Condition Specification
- Sweet Non-Chocolate Snacks (Other)
  Interventions: Other: Snack Condition Specification
- Dried Fruit (Other)
  Interventions: Other: Snack Condition Specification

INTERVENTIONS:
Other: Snack Condition Specification — Individuals recieve a different snack for every week of the study. This is viewed as 4 phases. Phase 1 measures of habitual chocolate candy consumption (1 week), Phase 2 assesses participants' chocolate consumption while anticipating an oncoming chocolate candy restriction (1 week), Phase 3 is the total chocolate candy restriction period, but participants will be given 3 non-chocolate-candy snack substitutes in a random order (1 week per snack type, 3 weeks total), and Phase 4 examines participants' chocolate candy consumption when the 3-week restriction is lifted (1 week).
  Other Names: Generic Branded Snack Foods (commerically available)

SUMMARY:
Craving differs from hunger because it occurs even when a person is in a satiated state and in the absence of an energy deficit. Craving is usually triggered by specific foods and may be attributable to certain sensory properties of foods. Foods that are craved are often regarded as less healthy choices, and are higher in energy content. Chocolate is one of the most commonly reported foods craved by people in this country. Together, craving for chocolate has been suggested to be a possible cause of weight gain and access to chocolate therefore needs to be restricted.

However, it remains unknown if restriction may induce maladaptive eating behaviors of chocolate cravers. The anticipation of going on a diet has been shown to cause restrained and disinhibited eaters to react by consuming more chocolate. In this study, we will examine if this response is also found in chocolate cravers when they are asked to undergo three weeks of chocolate restriction. This study will also examine chocolate cravers' response after the chocolate restriction is lifted. We hypothesize that chocolate consumption of cravers will increase both before and after chocolate restriction is imposed. We also hypothesize that chocolate craving is specific to the food rather than its sweet taste, and that chocolate cravers are less willing to substitute chocolate for salty snacks, natural snacks, and sweet non-chocolate snacks during the restriction.

ELIGIBILITY:
Inclusion Criteria:

Sixty adult participants (age 18-60 years) who are regular chocolate candy eaters (> 4 times/week, at least 1 serving each time) are needed to complete this study. Additional eligible criteria include:

* Subjects high and low in restraint/disinhibition based on TFEQ
* BMI between 18-35
* American born, or have lived in United States for majority of life, as different cultures have been shown to have lower chocolate preferences and consumption.
* Snack on a regular basis
* No allergies to test foods
* Not taking medications that affect appetite or metabolism
* Willing to comply to study protocol and to eat test meals
* Consume chocolate, or chocolate candies more than 4 times per week

Exclusion Criteria:

* If a participant does not fit the above requirements, they will be excluded from participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Intake in kcal | over one week at baseline and another week after chocolate restriction
  The primary objective of this study is to investigate the anticipatory- (before) and reactive-responses (after) of regular chocolate candy consumers to a three-week total chocolate candy restriction.

SECONDARY OUTCOMES:
Snack and Craving Preference | 6 weeks
  A secondary objective of this study is to examine if the observed responses before and after chocolate candy restriction can be predicted by participants' personality, ingestive behavior and food craving status. Providing different snacks to the participants during the restriction period will allow us to determine if craving is specific to specific foods, in the case of this study, chocolate. Cravings will be measured three times per week for six weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States